CLINICAL TRIAL: NCT04549558
Title: Multimodal Ultrasonographic Assessment of Ipsilateral Axillary Lymph Nodes in Patients With Breast Cancer: A STARD Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Ahmed Helmy, Resident doctor, Assiut University
Other Study IDs: AssiutU AAHelmy
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Multimodal Ultrasonographic Assessment of Axillary Lymph Nodes in Patients With Breast Cancer
Keywords: Strain Elastography, Grey-Scale Ultrasound, Carcinoma, Nodal, Axilla, Color-Doppler,
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal Ultrasound — Multimodal Ultrasound (Strain Ultrasound Elastography, Conventional Grey-Scale Ultrasound, Color-Doppler Ultrasound, and Ultrasound Guided Fine Needle Aspirate) on Axillary Lymph Nodes

SUMMARY:
Breast cancer (BrCa) is the most common malignant neoplasm in women worldwide with a continuous rise on both its incidence and cancer-related deaths. Accurate evaluation of the presence, extent and status (benign or malignant) of axillary lymph nodes (ALNs) in patients with BrCa has an important prognostic value, and is essential for disease staging and treatment planning. Many radiological diagnostic modalities have been utilized to assess the nature of ALNs in the pre-operative stage. Each modality has its weaknesses and strengths. Multimodal imaging combines two or more imaging modalities into one system to produce details in clinical diagnostic imaging that are more precise than any conventional imaging alone. Therefore, the present study is designed to assess the role of simultaneous multi-modal sonographic tools [conventional grey-scale ultrasound; US, Color-Doppler ultrasound; CDU, strain ultrasound elastography; UE) in evaluating the nature (benign or malignant) of ipsilateral ALNs in patients with primary BrCa together with comparing the diagnostic indices of each with that of all-together (combined modalities). A total of 30 patients with BrCa and US-visible ALNs will be included. All will be subjected to simultaneous examination by US, CDU, UE and US-guided FNA cytology examination of their ipsilateral ALNs. Data will be collected and analyzed using SPSS version 23. Area under the receiver Operating Characteristic (ROC) curve will be calculated and the diagnostic indices of each modality and of all modalities will be measured.

DETAILED DESCRIPTION:
BACKGROUND Breast cancer (BrCa) is the most common malignant neoplasm in women worldwide with a continuous rise on both its incidence and cancer-related deaths (1-3). Accurate evaluation of the presence, extent and status of axillary lymph nodes (ALNs) in patients with BrCa has an important prognostic value, and is essential for disease staging and treatment planning (4).

Historically, axillary lymph node dissection (ALND) and histopathology was used for staging BrCa, but with inevitable short- and long-term complications such as lymphedema, nerve injury, seroma and infection (5). Afterwards, sentinel lymph node (SLN) biopsy (SLNB) has gradually replaced ALND despite its invasive nature, unavoidable false negative results and post-operative complication, which are far less than those encountered with ALND (6). According to the American Society of Oncology Guidelines, If the SLNB results are negative, no further dissection is done because there is no survival benefit for performing ALND in this setting. Patients with positive SLNB results traditionally undergo "completion" ALND (6,7)

Grey-scale ultrasound (US) is a non-invasive method that plays an important role in the preoperative evaluation of ALNs and obtaining samples in patients with BrCa (8-11). Nevertheless, US is operator dependent and focuses mainly on the morphological features lymph nodes (LNs). Addition of Color-Doppler Ultrasound (CDU helps in assessing the presence and distribution of vasculature pattern as well as the resistive index (RI) of ALNs (11-13). Despite their promising results, US and CDU, studies showed very wide ranges and variations in sensitivity and specificity (8-13).

Real-time strain ultrasound elastography (UE) is an imaging technique that utilizes the long-established clinical concept that malignant lesions are often stiffer than normal tissues. The stiffness, a characteristic that can't be assessed by US nor CDU (14) and the UE has therefore been utilized to assess pathological changes in many organs, such as liver, breast, thyroid, muscle, Kidney, Prostate, and cervical LNs (Nicely reviewed in 14). Additionally, elastograms obtained by UE are color-coded images indicating differences in stiffness of portions of a target tissue. These color maps or images arise from analysis of the changes in the radiofrequency impulses before and after the rhythmic manual compression directed along the radiation axis. In addition, UE images are produced simultaneously with the conventional gray-scale US to ensure that images of the same node are precisely obtained (14). UE has also been used in assessing ALNs, but with variable and conflicting results (15,16). Two recent meta-analyses concluded that UE can provide additive useful information regarding ALN assessment prior to surgical procedure selection (17,18).

Other imaging modalities such as mammography, magnetic resonance imaging (MRI), multi-detector computed tomography (CT), Positron-emission tomography (PET-CT) were also tried, but their wide use is limited by their moderate sensitivity, low specificity, need for special protocol for ALNs assessment, law availability, high cost and radiation hazard (19-25).

Multimodal imaging combines two or more imaging modalities into one system to produce details in clinical diagnostic imaging that are more precise than any conventional imaging alone.

AIMS The present study is designed to assess the role of simultaneous multi-modal sonographic tools (US, CDU, UE) in evaluating the nature (benign or malignant) of ipsilateral ALNs in patients with primary BrCa together with comparing the diagnostic indices of each with that of all-together (combined modalities). In other words, whether adding UE to conventional grey-scale US and CDU will increase their diagnostic accuracy or not.

METHODS A: Type of the study: A prospective cohort diagnostic hospital-based study B: Study Setting: Department of Diagnostic Radiology, Assiut University Hospitals.

C: Sample Size Calculation: The study will include 30 consecutive patients with primary BrCa and ipsilateral ALNs of obscure nature visible by axillary conventional/grey-scale ultrasound (US) scan. In Each patient, one or more LN may be examined.

D: Study tools: All participants will be subjected to the following:

I. Screening clinical physical and Grey-scale ultrasound examination of the axilla With patients in the supine position, an experienced radiologist in conventional US, CDU, UE will perform the physical clinical examination using a Gray-scale digital US scanner (General Electric (GE, USA), equipped with a 7.5-13 MHz liner transducer will be performed first to assess for the presence of ALNs. Only the ipsilateral axillary region will be evaluated.

II. Conventional (grey-scale) ultrasound (US) Scoring of the ALNs A gray-scale conventional US scoring system of 5 criteria will be implemented. These include 1) Short-axis (S) diameter (S >7 mm = score 1; S ≤7 mm = score 0), 2) Long-to-short axis (L/S) diameter ratio (L/S; <2 = score 1; ≥ 2 = score 0), 3) The hilum long axis-to-node long axis (H/L) diameter ratio (H/L <0.5 = score 1; H/L ≥ 0.5 = score 0). 4) Border (irregular = score 1; regular =score 0), and 5) Cortical thickness (T >3 mm = score 1; T ≤ 3 mm = score 0). When the node did not have a hilar region, the cortical thickness will be regarded as ≥ 3 mm when the short-axis diameter is >3 mm (26) and Figure 2.

III. Color Doppler Ultrasound (CDU) examination of the ALNs After US, CDU will be performed as previously described (11-13) with the following precautions: 1) use of low wall filter and low velocity scale to be able to detect slow flow. 2) adjust color gain to maximum to help better blood flow demonstration and avoid noise artefacts. 3) place the transducer gently to avoid superficial vessels compression that may lead to an increase in vascular resistance. Intra-nodal blood flow in color Doppler studies will be classified into 4 categories: 1) central flow; 2) peripheral flow; or 3) Mixed peripheral and central, 4) absent flow. Central vessels are those appearing in both hilar and peri-hilar branches only. Peripheral vessels are those in the periphery that have no connection with the hilar vessel. Lymph nodes with both peripheral and central (mixed) flow will be grouped as mixed. If blood vessels are detected, 3 Doppler spectral waveforms will be obtained, and their mean will be calculated and considered as the resistivity index (RI). The RI is chosen as it is not dependent on the angle of insonation, and therefore, it can be accurately calculated even in small vessels. RI is calculated as follows: RI = Peak systolic velocity - end diastolic velocity/peak systolic velocity

IV. Strain ultrasound elastography (UE) of the ALNs UE images will be evaluated with a scoring system based on the percentage and distribution of the hypoechoic cortex regions with a visible hilum in ALN (Pattern I) or all the hypoechoic lymph nodes with an absent hilum (Pattern II).

In Pattern I (LN with Hila), scoring will be as follows (26):

1. the green portion occupied almost all of the cortex;
2. the blue portion occupies <50% of the cortex;
3. the blue portion occupies >50% of the cortex, with scattered the green portions;
4. the blue portion occupies almost all of the cortex;
5. the blue portion occupies almost all of the cortex, with a green ring on the edge of the node.

In pattern II (LN without Hila), scoring will be as follows (26):

1. Green portion occupying almost all of the cortex.
2. Blue portion occupying less than 50% of the cortex.
3. Blue portion occupying more than 50% of the cortex, with a scattered green portion
4. Blue portion occupying almost all of the cortex.
5. Blue portion occupying almost all of the cortex, with a green ring on the edge of the node.

Calculation of the Strain Ratio (SR) by UE. The SR is a ratio between the strain value of the two regions of interest (ROI) A and B, where ROI-A is the deepest blue portions of the hypoechoic regions within the nodes, and ROI-B is the surrounding soft and adipose tissue at the same depth.

(SR = strain value of ROI-B / strain value of ROI-A) Of note, SR is automatically calculated by the software built into certain equipment and displayed on its monitor (26).

V. Combined evaluation of gray-scale US, CDU and UE. The score of combined evaluation for each lymph node will be the sum of the gray-scale US (5 points), the CDU (1 point), and the UE (5 points) scores. A cut-off value will be evaluated with the pathological diagnosis.

VI. Ultrasound-guided FNA from the ALNs After completion of the above 3 sonographic modalities' examinations, and under local anesthesia using 5 ml of subcutaneous 1% Xylocaine, US-guided fine needle aspiration (FNA) will be performed by the same radiologist for all visible ALNs using 20-22 gauge needles attached to a 10 ml plastic syringe. Under UE guidance, the needle will be inserted into the cortex with 3 passes as routinely performed and previously described (27). When 2 or more abnormal LNs are identified, the node that looks the most suspicious will be aspirated. Samples will then be spread and fixed on glass-slides using 95% alcohol and air-dried for Pap & Diff-Quik (American Scientiﬁc Products, McGraw Park, IL, USA) staining in the Pathology Department prior to being examined. The final pathological diagnosis for the LNs will be made by a pathologist blinded to the imaging findings. Results of the US modalities will be correlated with the results of the FNAC.

E: Data Management and Statistical Analyses Data collection will be done in a preformed "Data Collection Form" (Appendix 1) prior to being entered in Microsoft Exel 2016. Afterwards, data will be exported to the Statistical Package for Social Sciences (SPSS) version 23.0 software package (SPSS, Inc., Chicago, IL, USA) for the statistical analysis. Comparisons of numeric (continuous) variables and categorical variables will be done using the Wilcoxon's rank sum test or Student's t-test and Chi-Square or Fisher's Exact test respectively and as appropriate. The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy will be calculated to compare the diagnostic performance of each modality. The areas under the receiver operating characteristic (ROC) curves (AUC) will be calculated and compared using the U-test. All cutoff values will be determined depending on the best accuracy identified by ROC curves. A probability value of (P<0.05) will be considered Statistically significant for all tests. The cytopathological diagnosis will be considered as the reference gold standard.

REFERENCES

1. Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019;69(1):7-34.
2. DeSantis CE, Ma J, Gaudet MM, et al. Breast cancer statistics, 2019. CA Cancer J Clin. 2019;69(6):438-451.
3. Bray F, Ferlay J, Soerjomataram I, et al. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin 2018;68:394-424.
4. Kleer CG, Sabel MS. Prognostic and predictive factors in breast cancer. In: Kuerer HM, ed. Kuerer's breast surgical oncology. New York, NY: McGrawHill, 2010; 244.
5. Ivens D, Hoe AL, Podd TJ, et al. Assessment of morbidity from complete axillary dissection. Br J Cancer 1992;66:136-138.
6. Lyman GH, Giuliano AE, Somerfield MR, et al. American Society of Clinical Oncology guideline recommendations for sentinel lymph node biopsy in early-stage breast cancer. J Clin Oncol. 2005;23(30):7703-7720.
7. Krag DN, Anderson SJ, Julian TB, et al. Technical outcomes of sentinel-lymph-node resection and conventional axillary-lymph-node dissection in patients with clinically node-negative breast cancer: results from the NSABP B-32 randomised phase III trial. Lancet Oncol 2007;8:881-888.
8. Britton, PD, Meroni S, Moscovici OC, et al. Use of ultrasound-guided axillary node core biopsy in staging of early breast cancer. Eur Radiol 2009;19:561-569.
9. Choi YJ, Ko EY, Han BK, et al. High-resolution ultrasonographic features of axillary lymph node metastasis in patients with breast cancer. Breast 2009;18:119-122.
10. Alvarez S, Añorbe E, Alcorta P, et al. Role of sonography in the diagnosis of axillary lymph node metastases in breast cancer: a systematic review. Am J Roentgenol 2006;186:1342-1348.
11. Choudhary J, Agrawal R, Mishra A, Nandwani R. Ultrasound and color Doppler evaluation of axillary lymph nodes in breast carcinoma with histopathological Correlation. Int J Scientific Study 2018;5(10):59-66.
12. Esen G, Gurses B, Yilmaz MH, et al. Gray scale and power Doppler US in the preoperative evaluation of axillary metastases in breast cancer patients with no palpable lymph nodes. Eur Radiol. 2005;15(6):1215-1223.
13. Esen G. Ultrasound of superficial lymph nodes. Eur J Radiol. 2006;58(3):345-359.
14. Sigrist RMS, Liau J, El Kaffas A, et al. Ultrasound Elastography: Review of Techniques and Clinical Applications. Theranostics 2017; 7:1303-1329.
15. Tsai WC, Lin CK, Wei HK, et al. Sonographic elastography improves the sensitivity and specificity of axilla sampling in breast cancer: a prospective study. Ultrasound Med Biol 2013;39:941-949.
16. Park YM, Fornage BD, Benveniste AP, et al. Strain elastography of abnormal axillary nodes in breast cancer patients does not improve diagnostic accuracy compared with conventional ultrasound alone. AJR Am J Roentgenol 2014;203(6):1371-1378.
17. Wang RY, Zhang YW, Gao ZM, Wang XM. Role of sonoelastography in assessment of axillary lymph nodes in breast cancer: a systematic review and meta-analysis. Clin Radiol 2020;75:320.e1-320.e7.
18. Tang GX, Xiao XY, Xu XL, et al. Diagnostic value of ultrasound elastography for differentiation of benign and malignant axillary lymph nodes: a meta-analysis. Clin Radiol 2020;75:481.e9-481.e16.
19. Valente SA, Levine GM, Silverstein MJ, et al. Accuracy of predicting axillary lymph node positivity by physical examination, mammography, ultrasonography, and magnetic resonance imaging. Ann Surg Oncol 2012;19:1825-1830.
20. Kim WH, Kim HJ, Lee SM, et al. Preoperative axillary nodal staging with ultrasound and magnetic resonance imaging: predictive values of quantitative and semantic features. Br J Radiol. 2018;91(1092):20180507.
21. Felipe VC, Graziano L, Barbosa PNVP, et al. Multidetector Computed Tomography with Dedicated Protocol for Breast Cancer Locoregional Staging: Feasibility Study. Diagnostics (Basel). 2020;10(7):479.
22. Liang X, Yu J, Wen B, et al. MRI and FDG-PET/CT based assessment of axillary lymph node metastasis in early breast cancer: a meta-analysis. Clin Radiol. 2017;72(4):295-301
23. Zhang X, Liu Y, Luo H, Zhang J. PET/CT and MRI for Identifying Axillary Lymph Node Metastases in Breast Cancer Patients: Systematic Review and Meta-Analysis [published online ahead of print, 2020 Jun 21]. J Magn Reson Imaging. 2020;10.1002/jmri.27246.
24. Marino MA, Avendano D, Zapata P, et al. Lymph node imaging in patients with primary breast cancer: concurrent diagnostic tools. The Oncologist 2020;25:e231-e242.
25. Lowes S, Leaver A, Cox K, et al. Evolving imaging techniques for staging axillary lymph nodes in breast cancer. Clin Radiol. 2018;73(4):396-409.
26. Xu Y, Bai X, Chen Y, et al. Application of Real-time Elastography Ultrasound in the Diagnosis of Axillary Lymph Node Metastasis in Breast Cancer Patients. Sci Rep. 2018;8(1):10234.
27. Krishnamurthy S, Sneige N, Bedi DG, et al. Role of ultrasound-guided fine-needle aspiration of indeterminate and suspicious axillary lymph nodes in the initial staging of breast carcinoma. Cancer. 2002;95(5):982-988.
28. https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/(Last seen on 25,8,2020).

ELIGIBILITY:
Inclusion Criteria:

Female patients with primary breast cancer (BrCa) and axillary lymph nodes (ALNs) referred to the Department of Diagnostic Radiology for pre-operative assessment of presence, extent and nature of ALNs.

Exclusion Criteria:

Patients with secondary or recurrent BrCa Patients exposed to loco-regional radio- or chemotherapy Patients with previous axilla surgery Presence of Distant metastasis (Liver, Bone, Lung) Patients who deny or refuse to participate in the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive female patients with primary breast cancer (BrCa) and axillary lymph nodes (ALNs) of unknown nature (benign or malignant) referred to the Department of Diagnostic Radiology for pre-operative assessment of presence, extent and nature of ALNs.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the role of Strain Elastography and other US modalities | 6-8 month
  Assessment of the role of multimodal ultrasonography in diagnosis/recognition of the nature of ALNs (benign or malignant) in patients with 1ry BrCa.

SECONDARY OUTCOMES:
Develop a Scoring system | 6-8 month
  Using the 4 modalities, a scoring system will be generated to predict the nature of ALNs (malignancy)

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] DeSantis CE, Ma J, Gaudet MM, Newman LA, Miller KD, Goding Sauer A, Jemal A, Siegel RL. Breast cancer statistics, 2019. CA Cancer J Clin. 2019 Nov;69(6):438-451. doi: 10.3322/caac.21583. Epub 2019 Oct 2. PMID 31577379
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593